CLINICAL TRIAL: NCT05261685
Title: Twelve-Month Outcome of Single-step Transepithelial Photorefractive Keratectomy for Moderate Hyperopia and Hyperopic Astigmatism
Brief Title: Single-step Transepithelial PRK for Hyperopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdel-Radi, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STEPRKH
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2022-07-12 (Actual); Status verified 2022-07

CONDITIONS: Moderate Hyperopia
Keywords: Single-step PRK; StreamLight PRK; Hyperopia; Photorefractive keratectomy
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hyperopic patients planned to undergo single-step transepithelial PRK (Experimental): Patients with moderate hyperopia or hyperopic astigmatism were planned to undergo transepithelial PRK using the new single-step StreamLight PRK Technology.
  Interventions: Procedure: Single-step transepithelial PRK

INTERVENTIONS:
Procedure: Single-step transepithelial PRK — Single-step transepithelial Photorefractive keratectomy (PRK) is a corneal refractive surgical procedure utilized to correct myopia, hyperopia and astigmatism where excimer laser is used in a single step to remove the corneal epithelium followed by stromal laser ablation to correct the patient's refractive error.

SUMMARY:
Hyperopia is one of the commonest refractive errors encountered in ophthalmology practice.

Laser in situ keratomileusis (LASIK) has been widely used to correct hyperopia especially with the advent of femtosecond laser technology allowing larger flap creation suitable for peripheral hyperopic ablations with resultant predictable, effective, and safe refractive outcomes. However, the encountered LASIK flap complications encouraged many surgeons to assess efficiency and safety of surface ablation techniques such as photorefractive keratectomy (PRK) to correct hyperopia.

DETAILED DESCRIPTION:
Although the initial refractive results of conventional manual or alcohol assisted PRK for hyperopia were encouraging, the frequently encountered post-PRK complications including undercorrection, overcorrection and regression of the hyperopic error had downgraded the conventional PRK as a preferred procedure for hyperopic correction.

Transepithelial PRK provides an alternative technique to uniformly remove the epithelium using the excimer laser to minimize the potential complications caused by mechanical or alcohol assisted epithelial removal in conventional PRK. Advances in transepithelial PRK technology have allowed refractive surgeons to remove the epithelium followed by stromal laser ablation in a single step instead of performing the procedure in 2 separate steps known as phototherapeutic keratectomy-photorefractive keratectomy (PTK-PRK).

Most of the previous studies paid particular attention to investigate the accuracy and safety of single-step transepithelial PRK in correcting myopia and myopic astigmatism. The aim of the current study is to evaluate the visual and refractive outcomes of the single-step transepithelial PRK procedure in correcting moderate hyperopia and hyperopic astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate hyperopia with a hyperopic cycloplegic spherical equivalent between +2 and + 4.5 diopters D.
* A steep keratometry (Ks) ≤ 46 D.
* Minimum pachymetry of 500 μm with a calculated residual stromal bed exceeding 350 μm after epithelial and stromal ablation.

Exclusion Criteria:

* Patients not candidate for corneal refractive surgery,
* Steep cornea (Ks > 46 D) with an expected postoperative keratometry > 48 D,
* Large angle kappa as estimated by Chord mu > 0.25 mm,
* Hyperopic amblyopia whether unilateral or bilateral with CDVA less than 0.2 . logMAR acuity,
* Recent contact lens wear, dry eye disease and autoimmune disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 12 months
  Uncorrected and corrected distance visual acuity (UDVA,CDVA) measurement using logMAR distant charts.
Cycloplegic refraction | 12 months
  Cycloplegic sphere, cylinder and refractive spherical equivalent (SEQ) were measured with auto-keratorefractometer (KR-8900:Topcon, Korea republic)

SECONDARY OUTCOMES:
Keratometry and corneal asphericity | 12 months
  Postoperative keratorefractive changes in mean keratometry (Km) and Q value were recorded using pentacam (Oculus GmbH, Germany)
Post-PRK haze | 12 months
  Post-PRK haze was evaluated using slit lamp based on Fantes et al. scale:
  Grade 0: No haze, completely clear cornea
  Grade 0.5: Trace haze seen with careful oblique illumination
  Grade 1: Haze not interfering with the visibility of fine details of the iris
  Grade 2: Mild obstruction of iris details
  Grade 3: Moderate obstruction of the iris and lens
  Grade 4: Complete opacification of the stroma in the area of the scar, anterior chamber is totally obscured.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Abdel-Radi, Principal Investigator — Assiut University
Locations (1):
- TIBA eye center, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adib-Moghaddam S, Arba-Mosquera S, Walter-Fincke R, Soleyman-Jahi S, Adili-Aghdam F. Transepithelial Photorefractive Keratectomy for Hyperopia: A 12-Month Bicentral Study. J Refract Surg. 2016 Mar;32(3):172-80. doi: 10.3928/1081597X-20160121-01. PMID 27027624
- [Derived] Abdel-Radi M, Rateb M, Saleh MGA, Aly MOM. Twelve-month outcomes of single-step transepithelial photorefractive keratectomy for moderate hyperopia and hyperopic astigmatism. Eye Vis (Lond). 2023 Mar 1;10(1):7. doi: 10.1186/s40662-023-00327-4. PMID 36855211